CLINICAL TRIAL: NCT01816035
Title: Thrombokinetic Studies of Ado-Trastuzumab Emtansine
Brief Title: Trastuzumab Emtansine in Treating Patients With HER2-Positive Metastatic or Locally Advanced Breast Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7900; NCI-2013-00552 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CC-7900; 7900 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: HER2/Neu Positive; Recurrent Breast Carcinoma; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (trastuzumab emtansine) (Experimental): Patients receive trastuzumab emtansine IV over 30-90 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving response may continue treatment.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Trastuzumab Emtansine

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Trastuzumab Emtansine — Given IV
  Other Names: Ado Trastuzumab Emtansine; Kadcyla; PRO132365; RO5304020; T-DM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate

SUMMARY:
This phase I trial studies the side effects and best way of giving trastuzumab emtansine in treating patients with human epidermal growth factor receptor 2 (HER2)-positive breast cancer that has spread to other parts of the body or nearby tissue and cannot be removed by surgery. Biological therapies, such as trastuzumab emtansine, may stimulate the immune system in different ways and stop cancer cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess change in thrombokinetics (platelet circulation life span).

SECONDARY OBJECTIVES:

I. Benefit rate (as defined by stable disease, partial response, or complete response by Response Evaluation Criteria in Solid Tumors [RECIST] v 1.1) at the end of study activities.

II. To evaluate the safety of trastuzumab emtansine (ado-trastuzumab emtansine) (non-platelet toxicity).

III. To evaluate the pharmacokinetics of ado-trastuzumab emtansine.

OUTLINE:

Patients receive trastuzumab emtansine intravenously (IV) over 30-90 minutes on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Patients achieving response may continue treatment.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Signed study-specific informed consent form
* Histologically or cytologically documented breast cancer
* Metastatic or unresectable locally advanced/recurrent breast cancer
* HER2-positive disease documented as in situ hybridization (ISH)-positive and/or 3+ by immunohistochemistry (IHC) on previously collected tumor tissue
* Absolute neutrophil count (ANC) > 1500 cells/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9.0 g/dL (patients are allowed to receive transfused red blood cells [RBC] to achieve this level)
* Total bilirubin =< 1.5 × upper limit of normal (ULN), except in patients with previously documented Gilbert's syndrome, in which case the direct bilirubin should be less than or equal to the ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 × ULN
* Alkaline phosphatase =< 2.5 × ULN (patients with hepatic and/or bone metastases: alkaline phosphatase =< 5 × ULN)
* Serum creatinine < 1.5 × ULN
* International normalized ratio (INR) < 1.5 × ULN
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Left ventricular ejection fraction (LVEF) >= 50% by either echocardiogram (ECHO) or multigated acquisition scan (MUGA)
* Negative results of serum pregnancy test for premenopausal women of reproductive capacity and for women < 12 months after entering menopause
* For women of childbearing potential and men with partners of childbearing potential, agreement by the patient and/or partner to use a highly effective, non-hormonal form of contraception or two effective forms of non-hormonal contraception; female patients of childbearing potential must agree to use two effective forms of non-hormonal contraception; effective methods of contraception include: intrauterine device (IUD); female condom; male condom; diaphragm with spermicide; cervical cap; or a sterile sexual partner; male patients with partners of childbearing potential must use barrier contraception; in addition, male patients should also have their partners use another method of contraception from the time of informed consent through the duration of study activity
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures, including thrombokinetic studies and platelet function studies

Exclusion Criteria:

CANCER-RELATED CRITERIA

* Known platelet disorder, such as von Willebrand's disease or baseline platelet count of < 100,000/mm^3
* Chemotherapy =< 21 days before first study treatment
* Trastuzumab =< 21 days before first study treatment
* Lapatinib =< 14 days before first study treatment
* Investigational therapy or any other therapy =< 28 days before first study treatment
* Any prior ado-trastuzumab emtansine
* Previous radiotherapy for the treatment of unresectable, locally advanced/recurrent or metastatic breast cancer is not allowed if:

  * The last fraction of radiotherapy has been administered within 14 days of first on-study thormbokinetic study
  * The patient has not recovered from any resulting acute toxicity (to grade =< 1) prior to first on-study thormbokinetic study
* Brain metastases that are untreated or symptomatic, or require any radiation, surgery, or steroid therapy to control symptoms from brain metastases within 14 days of first on-study thrombokinetic study; for patients with newly diagnosed brain metastases or unequivocal progression of brain metastases on screening scans, localized treatment (i.e., surgery, radiosurgery, and/or whole brain radiotherapy) is required before study enrollment; subjects with known brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 14 days of stable neurologic function prior to the first thrombokinetic procedure; patients with small brain metastases not symptomatic and deemed requiring treatment by managing clinicians or study investigators may be permitted to enroll on study
* History of intolerance (including grade 3 or 4 infusion reaction) or hypersensitivity to trastuzumab or murine proteins
* Current peripheral neuropathy of grade >= 3 per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.0
* Current use of any platelet functioning inhibitors (including aspirin) within 14 days of first on-study thrombokinetic study

CARDIOPULMONARY FUNCTION CRITERIA

* Current unstable ventricular arrhythmia requiring treatment
* History of symptomatic congestive heart failure (CHF) (New York Heart Association [NYHA] classes II-IV)
* History of myocardial infarction or unstable angina within 6 months of enrollment
* History of a decrease in LVEF to < 40% or symptomatic CHF with previous trastuzumab treatment
* Severe dyspnea at rest due to complications of advanced malignancy or requiring current continuous oxygen therapy

GENERAL CRITERIA

* Current severe, uncontrolled non-cancer systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease) resulting in a life expectancy of < 6 months
* Major surgical procedure or significant traumatic injury within 28 days before enrollment or anticipation of the need for major surgery during the course of study treatment
* Current pregnancy or lactation
* Current known active infection with human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C virus; for patients who are known carriers of hepatitis B virus (HBV), active hepatitis B infection must be ruled out based on negative serologic testing and/or determination of HBV deoxyribonucleic acid (DNA) viral load per local guidelines
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Platelet function, measured using a bleeding time test | Up to 30 days
Thrombokinetic changes | Baseline up to 30 days
  The actual analysis will fit a linear mixed effects model, using a two-sided Wald test to compare pre-therapy to the two post-therapy values, and should have greater power than a matched pairs design. Also, platelet lifespan may be measured in absolute terms (platelet lifespan) or relative terms (percentage relative to pre-therapy lifespan), and may be transformed to decrease the influence of extreme values.

SECONDARY OUTCOMES:
Cause of death | Up to 2 years
Clinical benefit rate | Up to 2 years
  Defined as the proportion of patients who achieve an objective response (complete response or stable disease) based on investigator assessment using Response Evaluation Criteria in Solid Tumors version 1.1 criteria at the conclusion of study procedures.
Death | Up to 2 years
Incidence of abnormal laboratory values | Up to 30 days after completion of study treatment
Incidence of adverse events leading to study treatment discontinuation, modification, or interruption, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after completion of study treatment
Incidence, type, and severity of adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after completion of study treatment
Incidence, type, and severity of severe adverse events graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after completion of study treatment
Left ventricular ejection fraction | Up to 2 years
Objective response rate, based on investigator assessment using Response Evaluation Criteria in Solid Tumors version 1.1 | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vijayakrishna Gadi, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States